CLINICAL TRIAL: NCT03616197
Title: The Effect Of Different Gingival Biotypes On Dimensional Stability Of Free Gingival Graft: A Comparative 6 Month Clinical Study
Brief Title: The Effect of Different Gingival Biotypes on Dimensional Stability of Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, serap karakış akcan, assistant professor doctor, Istanbul Aydın University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-9/7
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Gingival Recession; Atrophy
Keywords: gingival biotype of adjacent teeth; free gingival graft; shrinkage of graft
MeSH Terms: conditions — Gingival Recession; Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Determination of graft area measurements and shrinkage ratio of all photographs was performed by a periodontologist , an independent specialist who had not performed any surgical procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Thin Biotype group has described as Group 1. The biotypes of the terminal teeth adjacent to the free gingival graft region were determined by the "Probe transparency method".
  The mesial terminal tooth (MTT) was defined as the first tooth adjacent to the mesial side of the tooth / teeth to which the FGG will be applied. The distal terminal tooth (DTT) was defined as the first tooth adjacent to the distal side of the tooth / teeth to which the FGG will be applied. If MTT and DTT had thin biotype, the patient was assigned to the thin biotype group.
  Interventions: Procedure: free gingival graft
- Group 2 (Active Comparator): Thick biotype group has described as Group 2. The biotypes of the terminal teeth adjacent to the free gingival graft region were determined by the "Probe transparency method".
  The mesial terminal tooth (MTT) was defined as the first tooth adjacent to the mesial side of the tooth / teeth to which the FGG will be applied. The distal terminal tooth (DTT) was defined as the first tooth adjacent to the distal side of the tooth / teeth to which the FGG will be applied. If MTT and DTT had thick biotype, the patient was assigned to the thick biotype group.
  Interventions: Procedure: free gingival graft

INTERVENTIONS:
Procedure: free gingival graft — A horizontal incision was made along the mucogingival line with a scalpel number 15 to prepare a bed of periosteum and a thin immobilized connective tissue. The moving gingival tissues were removed coronally, and the bed was prepared so that the immobilized keratinized gingival tissue was preserved and the graft was placed apically. The template of the recipient region was placed in the donor region to be 2-3 mm more apically than the gingival margins of the teeth. The number of 15 scalpel was used to make incision at the template border and perpendicular to the keratinized tissue. The graft thickness was standardized in all patients between 1.5-2 mm. FGG was placed over the recipient bed and 5/0 non-resorbable monofilament sutures were used for fixing the four corners of the graft.

SUMMARY:
The aim of this study is to compare the effect of mesial and distal adjacent gingival biotypes of the tooth / teeth region of free gingival graft (FGG) on the shrinkage ratio of graft at 6 months postoperatively.

DETAILED DESCRIPTION:
The concept of gingival and periodontal phenotype was established as a result of clinical observation of changes in facial keratinized tissue width and thickness .It has been reported that gingival or periodontal diseases may develop more frequently in patients with thin gingival biotypes and that thick-flat biotype in implant restorations is important in achieving a successful aesthetic treatment outcome.

Free gingival graft (FGG) is a mucogingival surgical procedure that is successfully used in the presence of inadequate keratinized gingival width and gingival recession. It is thought that factors that may adversely affect the continuity of graft nutrition may be effective in graft shrinkage. These reasons can be listed as follows; graft thickness, traumatic surgical procedure, graft dehydration, and suturing procedure.

There was no study investigating the effect of periodontal biotypes on graft contraction in the region adjacent to the FGG operation.

ELIGIBILITY:
Inclusion Criteria:

* In the mandibular incisor tooth / teeth, the attached keratinized gingival width is <1 mm,
* No periodontal surgery has been performed previously on the involved tooth.
* In the absence of any systemic condition or illness (pregnancy, breastfeeding, mental retardation, diabetes, etc.) that may interfere with the patient's approval and dental treatment.
* Do not use any of the drug groups that may cause gingival overgrowth.

Exclusion Criteria:

* Previous periodontal surgery in the operation area
* Restoration of the buccal surface of the tooth and no pathology in the apical region of the tooth.
* In the presence of any systemic condition or illness (pregnancy, breastfeeding, mental retardation, diabetes, etc.) that may interfere with the patient's approval and dental treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The graft shrinkage ratio | baseline - 6th months postoperatively
  Graft shrinkage = Preoperative area - Postoperative area X 100 Preoperative area

SECONDARY OUTCOMES:
keratinized ginigival width | baseline - 6th months postoperatively
  Keratinized Gingival Width(KGW) was measured using a lugol solution (10% potassium iodide and 5% iodine) with a manual caliper spaced 0.5 mm from the mid-buccal point of the tooth, the distance between the gingival margin and mucogingival junction from MTT, DTT and the teeth/tooth in operation area.

CONTACTS AND LOCATIONS:
Overall Officials: serap karakış akcan, Phd, Study Director — İstanbul Aydın University, Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hatipoglu H, Keceli HG, Guncu GN, Sengun D, Tozum TF. Vertical and horizontal dimensional evaluation of free gingival grafts in the anterior mandible: a case report series. Clin Oral Investig. 2007 Jun;11(2):107-13. doi: 10.1007/s00784-006-0084-x. Epub 2007 Feb 9. PMID 17294229
- [Result] Gumus P, Buduneli E. Graft stabilization with cyanoacrylate decreases shrinkage of free gingival grafts. Aust Dent J. 2014 Mar;59(1):57-64. doi: 10.1111/adj.12149. Epub 2014 Feb 4. PMID 24494804
- [Result] Barbosa FI, Correa DS, Zenobio EG, Costa FO, Shibli JA. Dimensional changes between free gingival grafts fixed with ethyl cyanoacrylate and silk sutures. J Int Acad Periodontol. 2009 Apr;11(2):170-6. PMID 19431956